CLINICAL TRIAL: NCT06358872
Title: Azithromycine Pour la Vie Des Enfants au Niger II
Brief Title: Azithromycin for Child Survival in Niger II
Acronym: AVENIR II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de recherche et interventions en santé publique (CRISP) (Unknown); Ministère de la Santé Publique du Niger (Unknown); Le Programme National de Santé Oculaire (Unknown); Centre de Recherche Médicale et Sanitaire (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-39839
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Mortality; Antimicrobial Resistance
Keywords: Mass Treatment; Azithromycin; Childhood Mortality Rate; Antimicrobial Resistance; Implementation and Cost Analysis
MeSH Terms: interventions — Azithromycin; Suspensions

STUDY DESIGN:
Intervention Model Description: The intervention will involve biannual oral azithromycin MDA to children 1-59 months old distributed by community health workers. The Centre de Santé Integré (CSI) will be randomized to receive azithromycin MDA or delayed treatment in a stepped wedge design for the first 2 years. The delayed intervention arm will receive usual care for the first 2 years, then will receive the intervention for the next 2 years.
Who Masked: Outcomes Assessor
Masking Description: Participants, community health workers delivering the intervention, and team members supervising the program will not be masked. One biostatistician and one data analyst will remain unmasked to prepare the randomization sequence. Masked personnel include outcome assessors as well as the biostatistician and data analyst conducting the data analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Continuous Distribution (Active Comparator): Azithromycin distribution to children 1-59 months of age for four years using a door-to-door delivery approach via existing community health workers
  Interventions: Drug: Azithromycin for Oral Suspension
- Delayed Distribution (Active Comparator): Delayed, by two years, azithromycin distribution to children 1-59 months of age using a door-to-door delivery approach via existing community health workers
  Interventions: Drug: Azithromycin for Oral Suspension
- Stop Distribution (Active Comparator): Stopping azithromycin distribution after two years to children 1-59 months of age using a door-to-door delivery approach via existing community health workers
  Interventions: Drug: Azithromycin for Oral Suspension

INTERVENTIONS:
Drug: Azithromycin for Oral Suspension — Azithromycin will be administered as a single dose, in oral suspension form for children. The dose will be calculated by age or height depending on the child's age Both dosing cups and syringes will be used to administer treatment. For children too young to drink out of a dosing cup, a 1 ml or 5 ml syringe will be used, and the calculated dose will be rounded upwards to the nearest 0.2 ml.
  Other Names: Zithromax

SUMMARY:
Several randomized controlled trials have demonstrated that azithromycin mass drug administration (MDA) reduces child mortality, but increases antimicrobial resistance (AMR). The World Health Organization (WHO) guidelines for this intervention specify that implementation must be accompanied by continued monitoring of mortality and AMR. Niger is expanding the azithromycin MDA program nationwide. To establish monitoring of mortality and AMR as part of this program as well as to leverage the infrastructure to evaluate other child health interventions, AVENIR II is designed as an adaptive platform trial with monitoring and re-randomization every 2 years.

DETAILED DESCRIPTION:
AVENIR II is a cluster-randomized adaptive platform trial designed to evaluate community health interventions in Niger. The initial focus is to monitor under-5 mortality and antimicrobial resistance as the azithromycin MDA for child survival program expands in Niger, with the following specific aims:

1. Mortality.

   1. To conduct surveillance of mortality over time compared to the Sustainable Development Goal targets for under-5 mortality reduction. As this intervention is not intended to continue indefinitely, surveillance against a target is needed to determine when to stop.
   2. To continue to evaluate the effectiveness of azithromycin MDA to reduce under-5 mortality. Given the risk of AMR, the effectiveness of the intervention over time is needed to fully weigh the risks against the benefits.
2. Antimicrobial Resistance. To determine the impact of azithromycin MDA on AMR in population- and clinic-based samples.

ELIGIBILITY:
Inclusion Criteria:

CSI-level for mortality and AMR monitoring:

* Located in a region participating in the program
* Designated as rural by local study team
* Selected for participation in monitoring activities
* Safe and accessible for study teams
* Verbal approval from community leaders

Individual level for mortality monitoring:

* Residing in the catchment area of an eligible CSI
* Selected for participation in monitoring activities
* Female
* Age between 12 and 55 years old
* Verbal approval from participant

Individual-level for AMR monitoring:

* Residing in the catchment area of an eligible CSI
* Selected for participation in monitoring activities
* Age between 1 and 59 months old
* Verbal approval from a caregiver or guardian

Exclusion Criteria:

At the community-level:

* Designated as urban by local study team
* Inaccessible or unsafe for study team

At the individual-level:

* Known allergy to macrolides

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3300000 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2028-04-29 (Estimated); Study Completion 2028-04-29 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  Under-5 mortality rate (U5MR, deaths per 1,000 live births) assessed by pregnancy history at 2 years from the first treatment distribution, comparing the intervention and delayed arms
All-cause mortality | 4 years
  Under-5 mortality rate (U5MR, deaths per 1,000 live births) assessed by pregnancy history at 4 years, comparing the continue and stop arms
Prevalence of resistance to macrolides - nasopharyngeal swabs | 2 years
  Prevalence of macrolide-resistant pneumococcus from nasopharyngeal swabs in children 1-59 months old after 2 years of distributions, comparing the intervention and delayed arms
Prevalence of resistance to macrolides - nasopharyngeal swabs | 4 years
  Prevalence of macrolide-resistant pneumococcus from nasopharyngeal swabs in children 1-59 months old after 4 years of distributions, comparing the continue and stop arms
Load of genetic determinants of resistance to macrolides - rectal swabs | 2 years
  Load of genetic determinants of resistance to macrolides from rectal swabs in children 1-59 months old after 2 years of distributions, comparing the intervention and delayed arms
Load of genetic determinants of resistance to macrolides - rectal swabs | 4 years
  Load of genetic determinants of resistance to macrolides from rectal swabs in children 1-59 months old after 4 years of distributions, comparing the continue and stop arms

SECONDARY OUTCOMES:
Number of clinic visits - infectious | 2 years
  All infectious clinic visits among children 1-59 months of age in the program catchment area during the distribution period as assessed through passive surveillance of CSI records
Number of clinic visits - infectious | 4 years
  All infectious clinic visits among children 1-59 months of age in the program catchment area during the distribution period as assessed through passive surveillance of CSI records
Prevalence of Genetic Determinants of resistance - Nasopharyngeal swabs | 2 years
  Prevalence of genetic determinants of resistance from nasopharyngeal swabs in children 1-59 months old after 2 years of distributions, comparing the intervention and delayed arms
Prevalence of Genetic Determinants of resistance - Nasopharyngeal swabs | 4 years
  Prevalence of genetic determinants of resistance from nasopharyngeal swabs in children 1-59 months old after 4 years of distributions, comparing the continue and stop arms
Program Cost Per Dose Delivered | 2 years
  Program costs will be tracked using routine expenditure reporting and micro-costing activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran S O'Brien, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Program National de Santé Oculaire, Niamey, Niger

IPD SHARING:
Plan to Share IPD: Yes
De-identified data underlying outcomes publications will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication of the outcomes and will be made available indefinitely.
Access Criteria: Once made available, the data will be open access.

REFERENCES:
- [Background] Oldenburg CE, Ouattara M, Bountogo M, Boudo V, Ouedraogo T, Compaore G, Dah C, Zakane A, Coulibaly B, Bagagnan C, Hu H, O'Brien KS, Nyatigo F, Keenan JD, Doan T, Porco TC, Arnold BF, Lebas E, Sie A, Lietman TM. Mass Azithromycin Distribution to Prevent Child Mortality in Burkina Faso: The CHAT Randomized Clinical Trial. JAMA. 2024 Feb 13;331(6):482-490. doi: 10.1001/jama.2023.27393. PMID 38349371
- [Background] Sie A, Ouattara M, Bountogo M, Boudo V, Ouedraogo T, Compaore G, Dah C, Bagagnan C, Lebas E, Hu H, Rice J, Porco TC, Arnold BF, Lietman TM, Oldenburg CE. Azithromycin during Routine Well-Infant Visits to Prevent Death. N Engl J Med. 2024 Jan 18;390(3):221-229. doi: 10.1056/NEJMoa2309495. PMID 38231623
- [Background] Chao DL, Arzika AM, Abdou A, Maliki R, Karamba A, Galo N, Beidi D, Harouna N, Abarchi M, Root E, Mishra A, Lebas E, Arnold BF, Oldenburg CE, Keenan JD, Lietman TM, O'Brien KS. Distance to Health Centers and Effectiveness of Azithromycin Mass Administration for Children in Niger: A Secondary Analysis of the MORDOR Cluster Randomized Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2346840. doi: 10.1001/jamanetworkopen.2023.46840. PMID 38100110
- [Background] Keenan JD, Ayele B, Gebre T, Zerihun M, Zhou Z, House JI, Gaynor BD, Porco TC, Emerson PM, Lietman TM. Childhood mortality in a cohort treated with mass azithromycin for trachoma. Clin Infect Dis. 2011 Apr 1;52(7):883-8. doi: 10.1093/cid/cir069. PMID 21427395
- [Background] O'Brien KS, Cotter SY, Amza A, Kadri B, Nassirou B, Stoller NE, Zhou Z, West SK, Bailey RL, Keenan JD, Porco TC, Lietman TM. Childhood Mortality After Mass Distribution of Azithromycin: A Secondary Analysis of the PRET Cluster-randomized Trial in Niger. Pediatr Infect Dis J. 2018 Nov;37(11):1082-1086. doi: 10.1097/INF.0000000000001992. PMID 29561511
- [Background] Keenan JD, Bailey RL, West SK, Arzika AM, Hart J, Weaver J, Kalua K, Mrango Z, Ray KJ, Cook C, Lebas E, O'Brien KS, Emerson PM, Porco TC, Lietman TM; MORDOR Study Group. Azithromycin to Reduce Childhood Mortality in Sub-Saharan Africa. N Engl J Med. 2018 Apr 26;378(17):1583-1592. doi: 10.1056/NEJMoa1715474. PMID 29694816
- [Background] Doan T, Hinterwirth A, Worden L, Arzika AM, Maliki R, Abdou A, Kane S, Zhong L, Cummings ME, Sakar S, Chen C, Cook C, Lebas E, Chow ED, Nachamkin I, Porco TC, Keenan JD, Lietman TM. Gut microbiome alteration in MORDOR I: a community-randomized trial of mass azithromycin distribution. Nat Med. 2019 Sep;25(9):1370-1376. doi: 10.1038/s41591-019-0533-0. Epub 2019 Aug 12. PMID 31406349
- [Background] Keenan JD, Arzika AM, Maliki R, Elh Adamou S, Ibrahim F, Kiemago M, Galo NF, Lebas E, Cook C, Vanderschelden B, Bailey RL, West SK, Porco TC, Lietman TM; MORDOR-Niger Study Group. Cause-specific mortality of children younger than 5 years in communities receiving biannual mass azithromycin treatment in Niger: verbal autopsy results from a cluster-randomised controlled trial. Lancet Glob Health. 2020 Feb;8(2):e288-e295. doi: 10.1016/S2214-109X(19)30540-6. PMID 31981558
- [Background] WHO Guideline on Mass Drug Administration of Azithromycin to Children under Five Years of Age to Promote Child Survival [Internet]. Geneva: World Health Organization; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK561641/ PMID 32924384
- [Background] Doan T, Worden L, Hinterwirth A, Arzika AM, Maliki R, Abdou A, Zhong L, Chen C, Cook C, Lebas E, O'Brien KS, Oldenburg CE, Chow ED, Porco TC, Lipsitch M, Keenan JD, Lietman TM. Macrolide and Nonmacrolide Resistance with Mass Azithromycin Distribution. N Engl J Med. 2020 Nov 12;383(20):1941-1950. doi: 10.1056/NEJMoa2002606. PMID 33176084
- [Derived] Arzika AM, Amza A, Ousmane S, Maliki R, Almou I, Galo N, Harouna N, Mankara A, Aichatou B, Boubacar O, Lebas E, Peterson B, Brandt C, Picariello A, Cheng A, Porco TC, Doan T, Arnold BF, Lietman TM, O'Brien KS. Azithromycin mass drug administration to reduce child mortality in Niger (AVENIR II): a master protocol for a cluster-randomized adaptive platform trial to evaluate community-based health interventions. medRxiv [Preprint]. 2025 Jun 18:2025.06.17.25329431. doi: 10.1101/2025.06.17.25329431. PMID 40585143